CLINICAL TRIAL: NCT03077542
Title: Nonmyeloablative Haploidentical Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Sickle Cell Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 170069; 17-H-0069
Record Dates: First submitted 2017-03-10; First posted 2017-03-13 (Actual); Results first posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Sickle Cell Disease
Keywords: Peripheral Blood Stem Cells; Host-Donor Chimerism; Graft-Versus-Host Disease; Haploidentical; Donor Apheresis
MeSH Terms: conditions — Anemia, Sickle Cell; Graft vs Host Disease | interventions — Sirolimus; Alemtuzumab; Pentostatin; Cyclophosphamide; Hydroxyurea; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants (Experimental): Participants will receive pentostatin on days -21, -17, -13, and -9 and oral cyclophosphamide from days -21 to -8. Alemtuzumab to be infused on days -7 to -3, followed by 400 cGy TBI on day -1. Donor-derived peripheral blood stem cells will be given on Day 0 then cyclophosphamide will be given at 50 mg/kg on day +3. Sirolimus loading dose of 5mg PO q4h x three doses at one day after the completion of cyclophosphamide (on day +4) and continued the following day at 5mg PO q24h to maintain trough levels between 5-15 ng/ml.
  Interventions: Procedure: haploidentical stem cell transplant; Drug: Sirolimus; Drug: Alemtuzumab; Drug: Pentostatin; Drug: Cyclophosphamide; Drug: Hydroxyurea
- Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor (Other): A haploidentical relative donor will receive filgrastim (G-CSF) 10 to 16 µg/kg/d subcutaneously or intravenously for up to 6 days with apheresis collections of peripheral blood hematopoietic progenitor cells (PBPC) after the 5th day (and after the 6th day if required).
  Interventions: Drug: Filgrastim

INTERVENTIONS:
Procedure: haploidentical stem cell transplant — haploidentical stem cell transplant
  Arms: Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants
Drug: Sirolimus — conditioning regimen
  Other Names: Rapamune
  Arms: Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants
Drug: Alemtuzumab — conditioning regimen
  Other Names: Campth
  Arms: Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants
Drug: Pentostatin — conditioning regimen
  Other Names: Nipent
  Arms: Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants
Drug: Cyclophosphamide — conditioning regimen
  Other Names: Cytoxan
  Arms: Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants
Drug: Hydroxyurea — conditioning regimen
  Other Names: HU, Hydrea, Droxia
  Arms: Participants with Sickle Cell Disease with Nonmyeloablative Haplo Transplants
Drug: Filgrastim — A haploidentical relative donor will receive filgrastim (G-CSF) 10 to 16 µg/kg/d subcutaneously or intravenously for up to 6 days with apheresis collections of peripheral blood hematopoietic progenitor cells (PBPC) after the 5th day (and after the 6th day if required).
  Other Names: Granulocyte colony-stimulating factor (G-CSF)
  Arms: Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor

SUMMARY:
Background:

Peripheral blood stem cell transplantation procedures are used for people with sickle cell disease. Researchers want to improve the success and reduce the complications for these procedures. This might allow more people to have a transplant.

Objective:

To see if a new transplant regime is effective, safe and well tolerated in people with sickle cell disease.

Eligibility:

Adults at least 18 years old with sickle cell disease and certain complications.

A relative who is a half tissue match.

Design:

Participants will be screened with medical history, physical exam, and blood tests. Recipients will also have:

* Heart, lung, and mental health tests
* Chest x-rays
* Bone marrow taken from the pelvic bone
* Eyes and teeth checked

Recipients will have a large central line inserted into a vein for up to 6 months.

Donors will have their veins tested and have an IV inserted for 1 day or on rare occasions 2 days.

Donors will get a drug to activate bone marrow. It will be injected for about 6 days.

Donors will have at least 1 five-hour procedure where bone marrow stem cells will be collected. Blood will be taken from a vein in one arm or in rare cases from a groin vein and put through a machine. Some blood will be saved and the rest will be returned. Stem cells will be taken from the saved blood in a lab and frozen until ready to give to the recipient.

Recipients will have:

* Stems cells collected and frozen
* Hygiene lessons
* Bone density scans
* Low-dose radiation
* Drugs for their immune system
* Donor cells infused through their central line
* Transfusions

After about 30 days, recipients will leave the hospital. They must stay near NIH for 3 months after the transplant and have frequent visits. After returning home, they will have 8 visits over 5 years, then be contacted yearly.

DETAILED DESCRIPTION:
Nonmyeloablative allogeneic peripheral blood stem cell (PBSC) transplants are currently being investigated in phase I/II trials assessing engraftment, efficacy, and toxicity at a number of transplant centers. Our ongoing protocol for patients with severe congenital anemias, particularly sickle cell disease (SCD), and an HLA-matched sibling donor has had excellent preliminary results. None of the patients who engrafted had sickle-related events or any evidence of graft versus host disease (GVHD). There was no significant toxicity associated with the conditioning regimen. An additional protocol is ongoing for patients with high risk of graft rejection which employs pentostatin and oral cyclophosphamide (PC) pre-transplant to further deplete recipient lymphocytes in an attempt to decrease the rate of graft rejection. Four of 4 patients transplanted remain free of SCD.

Our main limitation has been a lack of HLA-matched sibling donors in the majority of patients. We performed a study in which patients with severe SCD who lacked a suitable donor underwent a search for a matched unrelated donor or umbilical cord donor. The vast majority of patients were not found to have an appropriate alternative donor. We therefore seek to develop a safe nonmyeloablative regimen to be applied to the haploidentical setting so that family members can serve as donors and greatly expand the donor pool.

We developed a nonmyeloablative haploidentical PBSC transplant protocol which included 3 cohorts, with stopping rules built in for regimen failure, defined as graft rejection or severe GVHD. All included 400 cGy total body irradiation (TBI) in divided doses 1 and 2 days prior to transplant, alemtuzumab, and sirolimus. The first cohort included no cyclophosphamide. The 2nd included one dose of cyclophosphamide given at 50mg/kg on day 3 post-transplant, and the 3rd included 100mg/kg cyclophosphamide given in divided doses on days 3 and 4 post-transplant. The engraftment rate and percentage of patients who remained free of SCD improved with each successive cohort. However, the graft rejection rate in the 3rd cohort remained high at 50%. To attempt to reduce the rate of graft rejection in the haploidentical setting, this protocol will add PC to the conditioning regimen.

In this protocol, we propose PBSC transplantation in patients with SCD considered at high risk for complications from or ineligible for standard bone marrow transplantation, with allogeneic peripheral blood stem cells from a haploidentical donor using a novel immunosuppressive regimen without myeloablation in an attempt to further decrease the transplant-related morbidity/mortality. The low intensity nonmyeloablative conditioning regimen will consist of a relatively low radiation dose for therapeutic radiation, Alemtuzumab (Campath ), Sirolimus (Rapamune ), Cyclophosphamide (Cytoxan ), and pentostatin (Nipent ) as a strategy to provide adequate immunosuppression to allow sufficient engraftment for clinical remission with a lower risk of GVHD development. T-cell replete, donor-derived, granulocyte colony-stimulating factor (G-CSF)- mobilized PBSC will be used to establish hematopoietic and lymphoid reconstitution.

The primary endpoint of this study is the percentage of patients at 100 days post-transplant who have not rejected their grafts, and who are without severe GVHD (defined as grade 3 and higher acute GVHD and moderate to severe chronic GVHD). Other endpoints include degree of donor-host chimerism necessary for long-term graft survival and disease amelioration, incidence of acute and chronic GVHD, incidence of graft rejection, transplant-related morbidity, as well as disease-free and overall survival.

ELIGIBILITY:
* INCLUSION CRITERIA-RECIPIENTS:

Patients with any type of sickle cell disease who are at high risk for disease-related cerebrovascular morbidity or early mortality, defined by having severe end-organ damage (A, B, C, D, or E):

A. A neurologic event resulting in focal neurologic deficits that lasted >= 24 hours (classical clinical definition of stroke, not requiring imaging studies of the brain) OR a focal neurological event resulting in abnormalities on T2- weighted or FLAIR images using an MRI scan, indicative of an acute infarct, with no other reasonable medical explanation (definition of a stroke supported with MRI imaging scans of the brain), OR both; OR

B. Tricuspid regurgitant jet velocity (TRV) of >= 2.7 m/s at baseline (without vaso- occlusive crisis) and/or pulmonary hypertension; OR

C. Sickle hepatopathy defined as either ferritin >1000 mcg/L and platelet count < 250,000/uL (without vaso-occlusive crisis) OR direct bilirubin > 0.4 mg/dL and platelet count <250,000/uL (without vaso- occlusive crisis)

D. Any acute chest syndrome episode resulting in intensive care admission requiring non- mechanical ventilatory support: simple nasal cannula, face mask that requires oxygen content (venti mask, non-rebreather), continuous positive airway pressure (CPAP), Bilevel positive airway pressure (BiPAP), high flow nasal cannula (HFNC) or invasive mechanical ventilatory support (delivered by endotracheal tube or tracheostomy).

E. Silent cerebral infarct defined as an infarct-like lesion based on an MRI signal abnormality at least 3 mm in one dimension and visible in two planes on FLAIR or T2- weighted images (or similar image with 3D imaging) and documented neurological examination performed by a neurologist demonstrating the participant has a normal neurologic or an abnormality on examination that could not be explained by the location of the brain lesion(s).

Non-disease specific:

A. Age greater than or equal to 18 years

B. Haploidentical relative donor available

C. Ability to comprehend and willing to sign an informed consent

D. Negative serum beta-HCG

E. Ejection fraction greater than or equal to 35%

F. Glomerular filtration rate >60 mL/min/1.73m^2 by cystatin C-based or iothalamate-based or other equivalent GFR testing

G. Adjusted DLCO greater than or equal to 35%

EXCLUSION CRITERIA RECIPIENT: (any of the following would exclude the subject from participating)

1. Available 6/6 HLA-matched sibling donor
2. ECOG performance status of 3 or more (See Appendix A)
3. Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen.
4. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.
5. Major anticipated illness or organ failure incompatible with survival from PBSC transplant
6. Pregnant or breast-feeding
7. Donor specific anti-HLA antibodies (DSAs) greater than or equal to 2000 Mean Fluorescence Intensity (MFI)
8. Patients seronegative for EBV who have EBV seropositive donors

INCLUSION CRITERIA-DONOR:

Haploidentical relative donor deemed suitable and eligible, and willing to donate, per clinical evaluations who are additionally willing to donate blood for research. Related donors will be evaluated in accordance with existing Standard NIH Policies and Procedures for determination of eligibility and suitability for clinical donation. Note that participation in this study is offered to all related donors, but is not required for a do le that not all related donors will enroll onto this study.

EXCLUSION CRITERIA-DONOR:

None

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2026-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney F Joseph, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-H-0069.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Sickle Cell Disease in Nonmyeloablative Haplo Blood Stem Cell Transplants: Participants will receive pentostatin on days -21, -17, -13, and -9 and oral cyclophosphamide from days -21 to -8. Alemtuzumab to be infused on days -7 to -3, followed by 400 cGy TBI on day -1. Donor derived peripheral blood stem cells will given on Day 0 then Cyclophosphamide will be given at 50 mg/kg on day +3. Sirolimus loading dose of 5mg PO q4h x three doses at one day after the completion of cyclophosphamide (on day +4) and continued the following day at 5mg PO q24h to maintain trough levels between 5-15 ng/ml.
Period: Overall Study
Arm/Group | Participants With Sickle Cell Disease in Nonmyeloablative Haplo Blood Stem Cell Transplants | Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor
Started | 28 | 29
Completed | 18 | 27
Not Completed | 10 | 2
Not completed — Death | 4 | 0
Not completed — Physician Decision | 6 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With Sickle Cell Disease With Nonmyeloablative Haplo Blood Stem Cell Transplants: Participants will receive pentostatin on days -21, -17, -13, and -9 and oral cyclophosphamide from days -21 to -8. Alemtuzumab to be infused on days -7 to -3, followed by 400 cGy TBI on day -1. Donor derived peripheral blood stem cells will be given on Day 0 then cyclophosphamide will be given at 50 mg/kg on day +3. Sirolimus loading dose of 5mg PO q4h x three doses at one day after the completion of cyclophosphamide (on day +4) and continued the following day at 5mg PO q24h to maintain trough levels between 5-15 ng/ml.
- Total: Total of all reporting groups
Arm/Group | Participants With Sickle Cell Disease With Nonmyeloablative Haplo Blood Stem Cell Transplants | Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 3 | 3
  Between 18 and 65 years | 28 | 26 | 54
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 13 | 14 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 28 | 55
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have Not Rejected Their Stem Cell Graft and Who Are Without Severe Graft-versus-host Disease Following Stem Cell Transplant
Description: The percentage of sickle cell participants at 100 days post-transplant who have not rejected their grafts and who are without severe graft-versus-host disease (GVHD). Severe GVHD is defined as grade 3 or higher for acute GVHD and moderate to severe for chronic GVHD according to NIH Consensus Criteria.
  Stem cell graft rejection is defined as
Time Frame: 100 days post transplant
Population: Analysis includes only those participants that received stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Sickle Cell Disease With Nonmyeloablative Haplo Blood Stem Cell Transplants
Number analyzed (Participants) | 22
Participants | 20

2. Secondary Outcome: Chimeric Value That is Required to Maintain Graft Survival and Hematologic Normalcy.
Description: The level of chimerism required to maintain both graft survival as well as hematologic normalcy. Hematologic normalcy may be defined as: being free from acute complications of sickle cell disease.
  The chimeric status of patients will be measured on days +14 (or when subject starts to engraft), +30, +60 and +100, and periodically after day +100, by microsatellite analysis of the peripheral blood.
  Engraftment of donor cells was assessed with the use of methods that detect informative polymorphisms in regions known to contain short tandem repeats. Peripheral-blood CD3+ T cells and CD14+CD15+ myeloid cells were selected for analysis with the use of immunomagnetic beads (Dynal).
Time Frame: Up to Year 5
Reporting Status: Not Posted

3. Secondary Outcome: Incidence of Donor Type Hemoglobin Post-transplant in SCD Patients Who Have Not Been Transfused in the Previous 3 Months.
Description: Incidence of donor type hemoglobin at 1 year post-transplant in SCD patients who have not been transfused in the previous 3 months.
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Number of Participants Who Developed Acute GVHD Grades I, II, III, IV
Description: Number of participants who developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grades are defined as:
  Grade I: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Day 100
Reporting Status: Not Posted

5. Secondary Outcome: Number of Participants Who Developed Moderate or Severe Chronic Graft vs Host Disease (GVHD)
Description: Number of Participants Who Developed Moderate or Severe Chronic Graft vs Host Disease (GVHD) up to 5 years.
  Moderate chronic GVHD involves EITHER 3 organs/sites with no clinically significant functional impairment OR a less than or equal to 1 organ/site with clinically significant functional impairment, but no major disability. Severe GVHD is associated with a major disability caused by chronic GVHD.
Time Frame: Up to Year 5
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participant That Are Disease-free Survival Following Stem Cell Transplant
Description: Percentage of participant that are disease-free survival following stem cell transplant. Disease-free survival is defined as alive and free acute complications related to sickle cell disease.
Time Frame: Up to Year 5
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Participant Overall Survival Following Stem Cell Transplant
Description: Percentage of Participant Overall Survival up to year 5 following stem cell transplant. Overall survival is defined as being alive following stem cell transplant.
Time Frame: Up to Year 5
Reporting Status: Not Posted

8. Secondary Outcome: Incidence of Graft Failure Following Stem Cell Transplant
Description: Incidence of graft failure following stem cell transplant. Graft failure is defined as the absence of or insufficient donor chimerism associated with the return of acute complications of sickle cell disease.
Time Frame: Up to 5 Years
Reporting Status: Not Posted

9. Secondary Outcome: Participant Graft Rejection Rate Following Stem Cell Transplant
Description: Participant graft rejection rate following stem cell transplant. Graft rejection is defined as donor myeloid chimerism and donor lymphoid chimerism <5%.
Time Frame: Up to 5 years
Reporting Status: Not Posted

10. Secondary Outcome: Number of Participants That Experienced Transplant-related Mortality
Description: Number of participants that experienced transplant-related mortality. Transplant-related mortality is defined as death that is at least possibly related to the transplant (GVHD, toxicity, infection, other causes).
Time Frame: 1 year
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants That Experienced Regimen Failure by Type of Haploidentical Donor
Description: Determine whether the type of haploidentical donor impacts the incidence of regimen failure. Number of participants that experienced regimen failure and type of haploidentical donor. Determine whether specific haploidentical donors (i.e. parent versus sibling versus child) will decrease the incidence of regimen failure. Haploidentical donor analyses include mother versus father, parent versus sibling, and parent versus child.
Time Frame: Up to Year 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse events will be collected from time of autologous stem cell collection/bone marrow harvest until completion of follow-up care post stem cell transplant. All AEs will be followed until satisfactory resolution.
Arm/Group | Participants With Sickle Cell Disease in Nonmyeloablative Haplo Blood Stem Cell Transplants | Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor
All-Cause Mortality (participants affected / at risk) | 4/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 25/28 | 1/29
Other Adverse Events (participants affected / at risk) | 26/28 | 2/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Sickle Cell Disease in Nonmyeloablative Haplo Blood Stem Cell Transplants (N=28) | Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor (N=29)
Anemia (Blood and lymphatic system disorders) | 6 (11) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Rapid ventricular response (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (7) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (5) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Unspecified Liver Lesion (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth infection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fall (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 7 (8) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 19 (97) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0)
Acute Graft versus Host Disease (aGVHD- GI) (Immune system disorders) | 1 (1) | 0 (0)
Angioedema (Immune system disorders) | 1 (1) | 0 (0)
Autoimmune hemolytic anemia (Immune system disorders) | 2 (2) | 0 (0)
Evans Syndrome (Immune system disorders) | 2 (2) | 0 (0)
Hemophagocytic Lymphohistiocytosis (HLH) (Immune system disorders) | 3 (3) | 0 (0)
Thrombotic-microangiopathy (TMA) (Immune system disorders) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 3 (3) | 0 (0)
Bacteremia (Infections and infestations) | 3 (3) | 0 (0)
CMV reactivation (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 infection (Infections and infestations) | 4 (4) | 0 (0)
EBV positive post-transplant lymphoproliferative disease (PTLD) (Infections and infestations) | 5 (5) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Influenza B (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
RSV infection (Infections and infestations) | 1 (1) | 0 (0)
Retropharyngeal fluid collection, + for Staph aureus (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Varicella zoster disease (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 4 (8) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Central apheresis line site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 8 (9) | 0 (0)
Platelet count decreased (Investigations) | 7 (7) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
SIADH (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (4) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Adverse drug reaction (Nervous system disorders) | 1 (1) | 0 (0)
Necrotizing leukoencephalopathy (Nervous system disorders) | 1 (2) | 0 (0)
Opioid toxicity (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (3) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (5) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Focal segmental glomerulosclerosis (FSGS) (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic Syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic range proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cryptogenic organizing pneumonia. (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Acute Skin Graft vs Host Disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Elective resection of seizure foci (Surgical and medical procedures) | 1 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 2 (3) | 0 (0)
Kidney biopsy (Surgical and medical procedures) | 2 (2) | 0 (0)
Splenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (4) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
Hemorrhagic shock (Vascular disorders) | 1 (1) | 0 (0)
Hypovolemic shock (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Sickle Cell Disease in Nonmyeloablative Haplo Blood Stem Cell Transplants (N=28) | Human Leukocyte Antigens (HLA) Haploidentical Related Stem Cell Donor (N=29)
Anemia (Blood and lymphatic system disorders) | 9 (19) | 0 (0)
Engraftment Syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 10 (12) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 18 (33) | 0 (0)
Suspected angioedema (Immune system disorders) | 1 (1) | 0 (0)
Vitiligo (Immune system disorders) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 3 (3) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 5 (7) | 0 (0)
CMV reactivation (Infections and infestations) | 7 (10) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Folliculitis/Furuncle (Infections and infestations) | 1 (1) | 0 (0)
Methicillin-susceptible Staphylococcus aureus (MSSA). (Infections and infestations) | 1 (1) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 6 (7) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 8 (11) | 0 (0)
Blood bilirubin increased (Investigations) | 8 (12) | 0 (0)
Febrile neutropenia (Investigations) | 1 (2) | 0 (0)
Hyperkalemia (Investigations) | 1 (1) | 0 (0)
Hypernatremia (Investigations) | 1 (3) | 0 (0)
Hyponatremia (Investigations) | 2 (2) | 0 (0)
Ferritin increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 16 (57) | 0 (0)
Neutrophil count decreased (Investigations) | 16 (61) | 2 (2)
Platelet count decreased (Investigations) | 11 (31) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 12 (44) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 4 (11) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Skin infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Serotonin syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (7) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eczematous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abscess aspiration (Surgical and medical procedures) | 1 (1) | 0 (0)
Splenectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-15): https://cdn.clinicaltrials.gov/large-docs/42/NCT03077542/Prot_SAP_000.pdf